CLINICAL TRIAL: NCT01462578
Title: Treatment of Patients With MDS or AML With an Impending Hematological Relapse With Azacitidine (Vidaza)
Brief Title: Treatment of Patients With Myelodysplastic Syndrome or Acute Myelocytic Leukemia With an Impending Hematological Relapse With Azacitidine (Vidaza)
Acronym: RELAZA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-RELA02-048; 2010-022388-37 (EudraCT Number); VZ-MDS-PI-0245 (Other: Celgene)
Record Dates: First submitted 2011-06-22; First posted 2011-10-31 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Acute Myelocytic Leukemia; Myelodysplastic Syndrome
Keywords: Neoplasms benign, malignant and unspecified; Acute myeloid leukemia; AML; Myelodysplastic syndrome; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neoplasms | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacytidine (Experimental): Azacytidine injection: 75 mg/m²/d, subcutaneous
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacytidine injection: 75 mg/m²/d, subcutaneous; initial minimum 6 cycles; another 6 or 12 cycles according to MRD niveau; maximum 24 cycles
  Other Names: Vidaza®

SUMMARY:
Assessment of efficacy of azacitidine to prevent a relapse

DETAILED DESCRIPTION:
Analysis of the effectiveness of azacitidine 6 months after start of therapy to prevent a hematological relapse in MDS or AML patients with significant residuals or an increase of minimal residual disease (MRD) which is defined as:

* decrease of CD34 donor chimerism (<80%) after allogeneic related or unrelated HSCT in CD34+ or CD117+ MDS or AML or
* increase in the AML-specific molecular markers in the quantitative PCR for t(6,9), NPM1+ AML >1% (ratio to reference gene) after conventional chemotherapy or allogeneic HSCT or
* persistence of the (above) MRD level >1% after conventional chemotherapy or allogeneic HSCT
* tolerance of azacitidine
* quality of the response of the MRD (major vs. minor) and the relapse-free survival and overall survival 12, 24 and 30 months after starting treatment with azacitidine
* modulation of CD34+, NK- and T-cells of MDS and AML patients by azacitidine

ELIGIBILITY:
Inclusion Criteria:

Screening:

* signed informed consent
* Age ≥18 years
* patients with MDS or AML after conventional chemotherapy or allogeneic HSCT and positive molecular marker such as t(6,9), NPM1 pos. or CD34+ or CD117+ in the case of an allogeneic HSCT

Treatment:

* MDS or AML without haematological relapse (blasts <5% in the bone marrow), and
* decrease of CD34 donor chimerism (<80%) after allogeneic related or unrelated HSCT in CD34+ or CD117+ MDS or AML or
* increase in the AML-specific molecular marker in the quantitative PCR for t(6,9), NPM1+ AML >1% after conventional chemotherapy or allogeneic HSCT or
* persistence of the (above) MRD levels >1% (relative to the reference gene) after conventional chemotherapy or allogeneic HSCT
* leukocytes > 3 Gpt/l and platelets >75 Gpt/l (transfusion independent)

Exclusion Criteria:

* Known history of hypersensitivity to any of the drugs used or their constituents or to drugs with similar chemical structure,
* Participation of the patient in another clinical trial within the last 4 weeks before the inclusion
* addiction or other disorders that do not allow the concerned person, to assess the nature and scope and possible consequences in the clinical investigation
* pregnant or breast feeding women
* women of childbearing potential, except women who meet the following criteria:

  * post-menopausal (12 months natural amenorrhea or 6 months amenorrhea with serum FSH >40 U/ml)
  * postoperative (6 weeks after hysterectomy with or without bilateral ovariectomy )
  * regular and proper use of a contraceptive method with error rate <1% per year (e.g., implants, depot injections, oral contraceptives, intrauterine device, IUD) during study treatment and up to 1 year after completion of therapy
  * sexual abstinence during study treatment and up to 1 year after completion of therapy
  * Vasectomy of the partner
* Men who do not use one of the following types of effective contraception during study treatment and up to 1 year after completion of therapy:

  * sexual abstinence
  * State post-vasectomy
  * Condom
* Evidence that the participating person is not expected to comply with the protocol (such as lack of cooperation)
* Uncontrolled active infection
* Severe hepatic impairment (AST and ALT may not exceed three times the normal) or liver cirrhosis or malignant liver tumor
* Dialysis dependent renal dysfunction
* Known severe congestive heart failure, incidence of clinically unstable cardiac or pulmonary disease These criteria are not for the screening phase up to a known allergic reaction to azacitidine or intolerance to apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-09; Primary Completion 2018-08 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with hematological relapse 6 months after start of treatment with azacitidin | 6 months after end of treatment

SECONDARY OUTCOMES:
Number of occurrence or exacerbation of clinical relevant acute or chronic GvHD | 2 years follow-up after treatment
Number of patients with infectious SAEs (rate of SAE) | 2 years follow-up after treatment
Rate of changes of methylation in CD34+ cells | 2 years follow-up after treatment
Relapse-free survival and overall survival | 12, 24 and 30 months after start of treatment
  Relapse-free survival and overall survival 12, 24 and 30 months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof. Dr., Principal Investigator — Universitätsklinikum Carl Gustav Carus, Medizinische Klinik und Poliklinik I, 01307 Dresden
Locations (11):
- Germany (11):
  - Charité Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Chemnitz (Küchwald), Chemnitz
  - Universitätsklinikum Carl Gustav Carus, Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Essen, Klinik für Hämatologie (Westdeutsches Tumorzentrum), Essen
  - Klinikum der J. W. Goethe-Universität, Medizinische Klinik II Hämatologie / Onkologie, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Medizinische Klinik, Abt. Innere Medizin V, Heidelberg
  - Klinikum rechts der Isar der TU München, III. Med. Klinik und Poliklinik, München
  - LMU München, Klinikum Großhadern, Med. Klinik III, München
  - Universitätsklinikum Münster, Innere Medizin A - KMT-Zentrum, Münster

REFERENCES:
- [Result] Platzbecker U, Middeke JM, Sockel K, Herbst R, Wolf D, Baldus CD, Oelschlagel U, Mutherig A, Fransecky L, Noppeney R, Bug G, Gotze KS, Kramer A, Bochtler T, Stelljes M, Groth C, Schubert A, Mende M, Stolzel F, Borkmann C, Kubasch AS, von Bonin M, Serve H, Hanel M, Duhrsen U, Schetelig J, Rollig C, Kramer M, Ehninger G, Bornhauser M, Thiede C. Measurable residual disease-guided treatment with azacitidine to prevent haematological relapse in patients with myelodysplastic syndrome and acute myeloid leukaemia (RELAZA2): an open-label, multicentre, phase 2 trial. Lancet Oncol. 2018 Dec;19(12):1668-1679. doi: 10.1016/S1470-2045(18)30580-1. Epub 2018 Nov 12. PMID 30442503
- [Derived] Platzbecker AS, Georgi JA, Middeke JM, Sockel K, Wehner R, Herbst RT, Wolf D, Baldus CD, Oelschlaegel U, Mutherig A, Fransecky L, Noppeney R, Bug G, Gotze KS, Kramer A, Bochtler T, Stelljes M, Esseling E, Stolzel F, von Bonin M, Serve H, Hanel M, Duhrsen U, Harig A, Muller-Tidow C, Schetelig J, Stasik S, Rollig C, Ehninger G, Kramer M, Schmitz M, Bornhauser M, Platzbecker U, Thiede C. Azacitidine to treat measurable residual disease in patients with MDS/AML: final long-term results of the RELAZA2 trial. Blood. 2025 Dec 8:blood.2025030816. doi: 10.1182/blood.2025030816. Online ahead of print. PMID 41359791
- See also: Website Study Alliance Leukemia (coordinating study group) — http://www.sal-aml.org